CLINICAL TRIAL: NCT04058665
Title: Hemostatic Agent Use and Intraoperative Blood Loss in Lumbar Spine Surgery
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: IRB00200167
Record Dates: First submitted 2019-08-14; First posted 2019-08-15 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2021-09

CONDITIONS: Blood Loss
Keywords: Lumbar spine surgery; Blood loss
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Observational group: No intervention performed. This is the overall group that will be retrospectively assessed for different variables pertaining to blood loss.
  Interventions: Device: Floseal

INTERVENTIONS:
Device: Floseal — Hemostatic agent

SUMMARY:
Perioperative variables that can be used to create a bundled approach quality improvement protocol to minimize blood loss in spine surgery will be evaluated using retrospective data collection and multivariate analysis of previously performed spinal surgeries at Johns Hopkins Hospital. In particular the investigators are interested in determining whether FloSeal® contributes towards increased control over perioperative bleeding compared to other hemostatic agents for potential inclusion in a future bundled approach.

DETAILED DESCRIPTION:
Blood loss is a major concern in spine surgery. Within lumbar fusion surgery, one study estimated an average blood loss of 800 mL (range 100-3,100 mL) for non-instrumented fusion and 1,517 mL (range 360-7,000 mL) for instrumented fusions. Blood transfusions are required in an estimated 8% to 36% of patients undergoing spine surgery.Transfusion promotes tissue perfusion and oxygen delivery during extensive surgeries, yet carries with it rare but significant risks. These include acute lung injury, febrile reactions, allergic episodes, infection, and impaired immune response. Given these potential risks, strategies to minimize extensive blood loss and resultant transfusion are warranted.

Previously described approaches in the literature that can minimize blood loss during spine surgery include: hypotensive anesthesia, hemostatic agents (e.g. FloSeal®), antifibrinolytic medications, advanced bipolar cautery (e.g. Aquamantys®), autologous blood salvage (e.g. Cell Saver®), perioperative and intraoperative temperature, operative time, nutritional state, coagulopathy, restrictive transfusion triggers, and rotational thromboelastometry (ROTEM).

Researchers in several medical fields have attempted to delineate comprehensive anemia prevention strategies described as "blood-saving bundles". A bundle encapsulates multiple evidence-based interventions that result in improved patient outcomes-here with a focus on reduced blood loss-when combined versus when each intervention is used in isolation. Care bundles applied to intensive care unit treatment and pneumonia, sepsis, and acute kidney injury care have demonstrated improved clinical outcomes. However, no bundled protocol currently exists that aim to decrease blood loss and transfusion incidence during spine surgery. Moreover, no data exist that identify whether use of FloSeal® over other hemostatic agents as part of a bundled protocol results in decreased blood loss and transfusion rates, improved surgical outcomes, and improved cost effectiveness.

Perioperative variables that can be used to create a bundled approach quality improvement protocol to minimize blood loss in spine surgery will be evaluated using retrospective data collection and multivariate analysis of previously performed spinal surgeries at Johns Hopkins Hospital. In particular the investigators are interested in determining whether FloSeal® contributes towards increased control over perioperative bleeding compared to other hemostatic agents for potential inclusion in a future bundled approach.

This retrospective multivariate analysis will identify potential factors associated with increased blood loss and transfusion incidence. The investigators anticipate using these findings to develop a future bundled protocol for implementation in all patients undergoing spine surgery at Johns Hopkins Hospital after approval by the Institutional Review Board. Such a bundled protocol has the potential to improve surgical outcomes and decrease institutional costs.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Undergoing lumbar spine surgery
* Surgery performed between July 1, 2016 and November 30, 2018
* Surgery performed at the Johns Hopkins East Baltimore Campus
* Available data on hemostatic agents used

Exclusion Criteria:

* Age under 18
* Surgery at location other than lumbar spine
* Surgical details unavailable
* Data unavailable for specified endpoints, including:

  * Hemostatic agent use
  * Blood loss
  * Operative time

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing lumbar spine surgery at Johns Hopkins Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Total blood loss | 1 week
  Cubic centimeters (cm^3) of blood loss throughout the operation.

SECONDARY OUTCOMES:
Length of hospital stay | Up to 1 month
  Days spent over entire hospital stay.
Number of postoperative infections | Up to 3 months
  All types of infection will be collected (surgical site infection, pneumonia, etc.)
Number of transfusion complications | Up to 1 month
  All possible transfusion complications
Number of medical complications | Up to 1 month
  Overall number of patient infections and transfusion complications.
Overall cost of care during time in hospital | Up to 1 year
  Total cost (dollars).
Operating room cost | Up to 1 year
  Cost (dollars) of the actual operation.
Total length of hospital stay cost | Up to 1 year
  Cost (dollars) included in the overall hospital stay.
Transfusion cost | Up to 1 year
  Cost (dollars) for the amount of transfusions the patient required.
Hospital disposition after surgery | Up to 1 month
  Postoperatively placed in the intensive care unit versus regular hospital floor.
Discharge disposition after surgery | Up to 1 month
  Discharged home versus discharged to a rehab facility.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Sciubba, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moller H, Hedlund R. Instrumented and noninstrumented posterolateral fusion in adult spondylolisthesis--a prospective randomized study: part 2. Spine (Phila Pa 1976). 2000 Jul 1;25(13):1716-21. doi: 10.1097/00007632-200007010-00017. PMID 10870149
- [Background] Berenholtz SM, Pronovost PJ, Mullany D, Garrett E, Ness PM, Dorman T, Klag MJ. Predictors of transfusion for spinal surgery in Maryland, 1997 to 2000. Transfusion. 2002 Feb;42(2):183-9. doi: 10.1046/j.1537-2995.2002.00034.x. PMID 11896333
- [Background] Butler JS, Burke JP, Dolan RT, Fitzpatrick P, O'Byrne JM, McCormack D, Synnott K, Poynton AR. Risk analysis of blood transfusion requirements in emergency and elective spinal surgery. Eur Spine J. 2011 May;20(5):753-8. doi: 10.1007/s00586-010-1500-0. Epub 2010 Jun 27. PMID 20582708
- [Background] Hu SS. Blood loss in adult spinal surgery. Eur Spine J. 2004 Oct;13 Suppl 1(Suppl 1):S3-5. doi: 10.1007/s00586-004-0753-x. Epub 2004 Jun 10. PMID 15197630
- [Background] Janssen SJ, Braun Y, Wood KB, Cha TD, Schwab JH. Allogeneic blood transfusions and postoperative infections after lumbar spine surgery. Spine J. 2015 May 1;15(5):901-9. doi: 10.1016/j.spinee.2015.02.010. Epub 2015 Feb 11. PMID 25681582
- [Background] Nuttall GA, Horlocker TT, Santrach PJ, Oliver WC Jr, Dekutoski MB, Bryant S. Predictors of blood transfusions in spinal instrumentation and fusion surgery. Spine (Phila Pa 1976). 2000 Mar 1;25(5):596-601. doi: 10.1097/00007632-200003010-00010. PMID 10749636
- [Background] Blajchman MA, Dzik S, Vamvakas EC, Sweeney J, Snyder EL. Clinical and molecular basis of transfusion-induced immunomodulation: summary of the proceedings of a state-of-the-art conference. Transfus Med Rev. 2001 Apr;15(2):108-35. doi: 10.1053/tmrv.2001.22614. No abstract available. PMID 11309732
- [Background] Burrows L, Tartter P. Effect of blood transfusions on colonic malignancy recurrent rate. Lancet. 1982 Sep 18;2(8299):662. doi: 10.1016/s0140-6736(82)92764-7. No abstract available. PMID 6125797
- [Background] Cannon RM, Brown RE, St Hill CR, Dunki-Jacobs E, Martin RC 2nd, McMasters KM, Scoggins CR. Negative effects of transfused blood components after hepatectomy for metastatic colorectal cancer. Am Surg. 2013 Jan;79(1):35-9. PMID 23317602
- [Background] de Almeida JP, Vincent JL, Galas FR, de Almeida EP, Fukushima JT, Osawa EA, Bergamin F, Park CL, Nakamura RE, Fonseca SM, Cutait G, Alves JI, Bazan M, Vieira S, Sandrini AC, Palomba H, Ribeiro U Jr, Crippa A, Dalloglio M, Diz Mdel P, Kalil Filho R, Auler JO Jr, Rhodes A, Hajjar LA. Transfusion requirements in surgical oncology patients: a prospective, randomized controlled trial. Anesthesiology. 2015 Jan;122(1):29-38. doi: 10.1097/ALN.0000000000000511. PMID 25401417
- [Background] Engoren MC, Habib RH, Zacharias A, Schwann TA, Riordan CJ, Durham SJ. Effect of blood transfusion on long-term survival after cardiac operation. Ann Thorac Surg. 2002 Oct;74(4):1180-6. doi: 10.1016/s0003-4975(02)03766-9. PMID 12400765
- [Background] Gilliss BM, Looney MR, Gropper MA. Reducing noninfectious risks of blood transfusion. Anesthesiology. 2011 Sep;115(3):635-49. doi: 10.1097/ALN.0b013e31822a22d9. PMID 21792054
- [Background] Glance LG, Dick AW, Mukamel DB, Fleming FJ, Zollo RA, Wissler R, Salloum R, Meredith UW, Osler TM. Association between intraoperative blood transfusion and mortality and morbidity in patients undergoing noncardiac surgery. Anesthesiology. 2011 Feb;114(2):283-92. doi: 10.1097/ALN.0b013e3182054d06. PMID 21239971
- [Background] Koch CG, Li L, Duncan AI, Mihaljevic T, Loop FD, Starr NJ, Blackstone EH. Transfusion in coronary artery bypass grafting is associated with reduced long-term survival. Ann Thorac Surg. 2006 May;81(5):1650-7. doi: 10.1016/j.athoracsur.2005.12.037. PMID 16631651
- [Background] Kuduvalli M, Oo AY, Newall N, Grayson AD, Jackson M, Desmond MJ, Fabri BM, Rashid A. Effect of peri-operative red blood cell transfusion on 30-day and 1-year mortality following coronary artery bypass surgery. Eur J Cardiothorac Surg. 2005 Apr;27(4):592-8. doi: 10.1016/j.ejcts.2005.01.030. PMID 15784356
- [Background] Popovsky MA. Transfusion-related acute lung injury: three decades of progress but miles to go before we sleep. Transfusion. 2015 May;55(5):930-4. doi: 10.1111/trf.13064. No abstract available. PMID 25959215
- [Background] Roberson RS, Bennett-Guerrero E. Impact of red blood cell transfusion on global and regional measures of oxygenation. Mt Sinai J Med. 2012 Jan-Feb;79(1):66-74. doi: 10.1002/msj.21284. PMID 22238040
- [Background] Ross A, Mohammed S, Vanburen G, Silberfein EJ, Artinyan A, Hodges SE, Fisher WE. An assessment of the necessity of transfusion during pancreatoduodenectomy. Surgery. 2013 Sep;154(3):504-11. doi: 10.1016/j.surg.2013.06.012. PMID 23972656
- [Background] Vamvakas EC, Blajchman MA. Transfusion-related mortality: the ongoing risks of allogeneic blood transfusion and the available strategies for their prevention. Blood. 2009 Apr 9;113(15):3406-17. doi: 10.1182/blood-2008-10-167643. Epub 2009 Feb 2. PMID 19188662
- [Background] Dutton RP. Controlled hypotension for spinal surgery. Eur Spine J. 2004 Oct;13 Suppl 1(Suppl 1):S66-71. doi: 10.1007/s00586-004-0756-7. Epub 2004 Jun 9. PMID 15197633
- [Background] Paul JE, Ling E, Lalonde C, Thabane L. Deliberate hypotension in orthopedic surgery reduces blood loss and transfusion requirements: a meta-analysis of randomized controlled trials. Can J Anaesth. 2007 Oct;54(10):799-810. doi: 10.1007/BF03021707. PMID 17934161
- [Background] Baird EO, McAnany SJ, Lu Y, Overley SC, Qureshi SA. Hemostatic Agents in Spine Surgery: A Critical Analysis Review. JBJS Rev. 2015 Jan 13;3(1):e2. doi: 10.2106/JBJS.RVW.N.00027. No abstract available. PMID 27501022
- [Background] Alvarez JC, Santiveri FX, Ramos I, Vela E, Puig L, Escolano F. Tranexamic acid reduces blood transfusion in total knee arthroplasty even when a blood conservation program is applied. Transfusion. 2008 Mar;48(3):519-25. doi: 10.1111/j.1537-2995.2007.01564.x. Epub 2007 Dec 7. PMID 18067499
- [Background] Frank SM, Wasey JO, Dwyer IM, Gokaslan ZL, Ness PM, Kebaish KM. Radiofrequency bipolar hemostatic sealer reduces blood loss, transfusion requirements, and cost for patients undergoing multilevel spinal fusion surgery: a case control study. J Orthop Surg Res. 2014 Jul 5;9:50. doi: 10.1186/s13018-014-0050-2. PMID 24997589
- [Background] Williamson KR, Taswell HF. Indications for intraoperative blood salvage. J Clin Apher. 1990;5(2):100-3. PMID 2404968
- [Background] Waters JH, Ness PM. Patient blood management: a growing challenge and opportunity. Transfusion. 2011 May;51(5):902-3. doi: 10.1111/j.1537-2995.2011.03122.x. No abstract available. PMID 21545588
- [Background] Manjuladevi M, Vasudeva Upadhyaya K. Perioperative blood management. Indian J Anaesth. 2014 Sep;58(5):573-80. doi: 10.4103/0019-5049.144658. PMID 25535419
- [Background] Carless PA, Henry DA, Carson JL, Hebert PP, McClelland B, Ker K. Transfusion thresholds and other strategies for guiding allogeneic red blood cell transfusion. Cochrane Database Syst Rev. 2010 Oct 6;(10):CD002042. doi: 10.1002/14651858.CD002042.pub2. PMID 20927728
- [Background] Carson JL, Terrin ML, Noveck H, Sanders DW, Chaitman BR, Rhoads GG, Nemo G, Dragert K, Beaupre L, Hildebrand K, Macaulay W, Lewis C, Cook DR, Dobbin G, Zakriya KJ, Apple FS, Horney RA, Magaziner J; FOCUS Investigators. Liberal or restrictive transfusion in high-risk patients after hip surgery. N Engl J Med. 2011 Dec 29;365(26):2453-62. doi: 10.1056/NEJMoa1012452. Epub 2011 Dec 14. PMID 22168590
- [Background] Hajjar LA, Vincent JL, Galas FR, Nakamura RE, Silva CM, Santos MH, Fukushima J, Kalil Filho R, Sierra DB, Lopes NH, Mauad T, Roquim AC, Sundin MR, Leao WC, Almeida JP, Pomerantzeff PM, Dallan LO, Jatene FB, Stolf NA, Auler JO Jr. Transfusion requirements after cardiac surgery: the TRACS randomized controlled trial. JAMA. 2010 Oct 13;304(14):1559-67. doi: 10.1001/jama.2010.1446. PMID 20940381
- [Background] Hebert PC, Wells G, Blajchman MA, Marshall J, Martin C, Pagliarello G, Tweeddale M, Schweitzer I, Yetisir E. A multicenter, randomized, controlled clinical trial of transfusion requirements in critical care. Transfusion Requirements in Critical Care Investigators, Canadian Critical Care Trials Group. N Engl J Med. 1999 Feb 11;340(6):409-17. doi: 10.1056/NEJM199902113400601. PMID 9971864
- [Background] Naik BI, Pajewski TN, Bogdonoff DI, Zuo Z, Clark P, Terkawi AS, Durieux ME, Shaffrey CI, Nemergut EC. Rotational thromboelastometry-guided blood product management in major spine surgery. J Neurosurg Spine. 2015 Aug;23(2):239-49. doi: 10.3171/2014.12.SPINE14620. Epub 2015 May 22. PMID 26053893
- [Background] Riessen R, Behmenburg M, Blumenstock G, Guenon D, Enkel S, Schafer R, Haap M. A Simple "Blood-Saving Bundle" Reduces Diagnostic Blood Loss and the Transfusion Rate in Mechanically Ventilated Patients. PLoS One. 2015 Sep 30;10(9):e0138879. doi: 10.1371/journal.pone.0138879. eCollection 2015. PMID 26421920
- [Background] Meybohm P, Richards T, Isbister J, Hofmann A, Shander A, Goodnough LT, Munoz M, Gombotz H, Weber CF, Choorapoikayil S, Spahn DR, Zacharowski K. Patient Blood Management Bundles to Facilitate Implementation. Transfus Med Rev. 2017 Jan;31(1):62-71. doi: 10.1016/j.tmrv.2016.05.012. Epub 2016 May 28. PMID 27317382
- [Background] Bagshaw SM. Acute Kidney Injury Care Bundles. Nephron. 2015;131(4):247-51. doi: 10.1159/000437152. Epub 2015 Dec 17. PMID 26673455
- [Background] Black MD, Vigorito MC, Curtis JR, Phillips GS, Martin EW, McNicoll L, Rochon T, Ross S, Levy MM. A multifaceted intervention to improve compliance with process measures for ICU clinician communication with ICU patients and families. Crit Care Med. 2013 Oct;41(10):2275-83. doi: 10.1097/CCM.0b013e3182982671. PMID 24060769
- [Background] Levy MM, Rhodes A, Phillips GS, Townsend SR, Schorr CA, Beale R, Osborn T, Lemeshow S, Chiche JD, Artigas A, Dellinger RP. Surviving Sepsis Campaign: association between performance metrics and outcomes in a 7.5-year study. Crit Care Med. 2015 Jan;43(1):3-12. doi: 10.1097/CCM.0000000000000723. PMID 25275252
- [Background] Lim WS, Rodrigo C, Turner AM, Welham S, Calvert JM; British Thoracic Society. British Thoracic Society community-acquired pneumonia care bundle: results of a national implementation project. Thorax. 2016 Mar;71(3):288-90. doi: 10.1136/thoraxjnl-2015-206834. Epub 2015 Jul 21. PMID 26197815